CLINICAL TRIAL: NCT04021680
Title: Far Eastern Memorial Hospital
Brief Title: Clinical Effectiveness of First Trimester Pre-eclampsia Screening Program.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Head of Department of Obstetrics & Gynecology, Associate Professor, Far Eastern Memorial Hospital
Other Study IDs: 108051-F
Record Dates: First submitted 2019-07-14; First posted 2019-07-16 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pre-eclampsia screening program — This screening program included the use of ultrasound, biomarkers and maternal factors in calculating the risk of developing preeclampsia.

SUMMARY:
To evaluate the clinical effectiveness of this screening program in preventing pre-eclampsia.

DETAILED DESCRIPTION:
The incidence of pre-eclampsia is about 2-8%, it is a leading cause of maternal and perinatal mortality and morbidity. Both ACOG (American Congress of Obstetricians and Gynecologists) and NICE (National Institute for Health and Clinical Excellence) guideline advocate the use of traditional screening method, which uses demographic characters and medical history to identify high risk women. This method detects only 35-40% of pre-eclampsia women. Study has shown that combination of maternal factors and biomarkers (uterine artery pulsatility index, placenta growth factor, PlGF; pregnancy associated plasma protein-A, PAPP-A) improves the detection rate.

In Taiwan, the prevalence of pre-eclampsia is about 1.21%. The incidence of pre-eclampsia is correlated with maternal age, with a relative risk of 5.13-fold in women aged 40 and above. Marrying late predisposes these women at high risk of developing pre-eclampsia. Our institution will be implementing first-trimester screening program starting from April 2019, this study aims to evaluate the clinical effectiveness of this screening program in preventing pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

- Women who are 20 years of age or older with singleton pregnancy between 11 to 13 + 6 weeks and received first trimester pre-eclampsia screening test in this institution.

Exclusion Criteria:

* Women who are not regularly inspected or not receiving prenatal care in this institution.
* Women who received first trimester pre-eclampsia screening test at other institution

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant woman
Study Population: women with with singleton pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of this screening program to detect preeclampsia | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No